CLINICAL TRIAL: NCT02705742
Title: Efficacy of Adipose Tissue Derived Autologous Repeated Mesenchymal Stem Cells Transplantation Via Hepatic Artery and Peripheral Vein in Patients With Liver Cirrhosis Due to HCV Hepatitis
Brief Title: Mesenchymal Stem Cells Transplantation for Liver Cirrhosis Due to HCV Hepatitis
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Saglik Bilimleri Universitesi Gulhane Tip Fakultesi (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GMMA-HCV-MSC-1
Record Dates: First submitted 2016-03-07; First posted 2016-03-10 (Estimated); Last update posted 2016-06-07 (Estimated); Status verified 2016-06

CONDITIONS: Liver Cirrhosis
Keywords: Mesenchymal stem cells; Liver cirrhosis; Hepatitis C
MeSH Terms: conditions — Liver Cirrhosis; Hepatitis C

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- stem cells group (Other): mesenchymal stem cells only
  Interventions: Biological: Mesenchymal Stem Cells

INTERVENTIONS:
Biological: Mesenchymal Stem Cells — 1.000.000 (one million) cells/kg, IV of dose in the Peripheral vein and 3.000.000 (three million) cells/kg of dose into the right hepatic artery)

SUMMARY:
In this study, investigators aimed to transplant autologous, adipose tissue derived mesenchymal stem cells to the patients with liver cirrhosis due to HCV. We also aimed to assess liver tissue regeneration, downgrade of clinical findings and antiviral efficacy. Finally investigators aimed to establish an alternative treatment modality to liver transplantation.

DETAILED DESCRIPTION:
In this study, investigators aimed to transplant autologous, adipose tissue derived mesenchymal stem cells to the patients with liver cirrhosis. Investigators also aimed to assess liver tissue regeneration, downgrade of clinical findings and antiviral efficacy. Finally investigators aimed to establish an alternative treatment modality to liver transplantation.

Hepatitis C Virus (HCV) which can lead to chronic hepatitis, liver cirrhosis and hepatocellular carcinoma (HCC) is an important health problem especially in western countries. In 5% - 25 of patients with chronic HCV hepatitis who are nonresponders to current medical treatment, liver cirrhosis develops. Approximately 1/3 of patients with liver cirrhosis become decompensate in 10 years. Medical treatment of liver cirrhosis, the last stage of the illness that leads to morbidity and mortality is difficult. Liver transplantation is still the most effective treatment for the patients with liver cirrhosis due to chronic hepatitis C, However, serious problems are accompanied with liver transplantation. Lack of liver donors, complications during and after the surgery, graft rejection and high costs are the main problems.

There are cells in the human body that are capable to renew themselves and differentiate to a diverse range of specialized cell types. These are called "stem cells". Stem cells can be differentiated to specialized cells in appropriate medias in the laboratory. Recently, the differentiation potential of mesenchymal stem cells (MSCs) into hepatocytes is proved by demonstrating hepatocytes containing Y chromosome in the female who has had bone marrow transplantation from male donors. In many laboratory studies, it is observed that human adipose tissue derived mesenchymal stem cells, transplanted to animals with induced liver damage, differentiate into the albumin producing hepatocytes. Even though the number of studies on human for the same purpose is few, findings are supporting those of animal experiments. Some very recent studies emphasize the antiviral effects of MSCs. The reasons for choosing this study title is; no available medical treatment for the non-responder cirrhotic patients, shortage of organ donors, patients rapidly progressing to transplantation candidates, and patients dying while they are in waiting lists and finally hopeful data regarding MSC applications. This is a hopeful, avant garde and sophisticated study which may constitute new horizons in context of cellular therapies.

In this study autologous adipose tissue derived MSCs will be transplanted to patients with liver cirrhosis due to chronic hepatitis C. After invitro expansion, patients will receive 1 million cells per kg. via peripheral vein every week for 3 times. Also via hepatic artery, 3 million cells per kg will be infused for 3 times in every 2 weeks. With this protocol, investigators aimed to increase liver regeneration, decrease in liver fibrosis, increase the waiting time of patients in transplantation lists and finally to establish a new and regenerative treatment protocol alternative to liver transplantation. For observation of clinical and laboratory improvement, patients are planned to be monitored by pathology examination of liver biopsies before and at 6th month after the treatment, monthly biochemical and hematologic blood tests and periodic radiologic examinations.

ELIGIBILITY:
Inclusion Criteria:

* Clinical, radiologic and pathologically proven Liver Cirrhosis Due to HCV Hepatitis
* Patients with no hepatic malignancies
* No co-existing serious respiratory and/or cardiovascular morbidities
* Patients who approved to join the study group with informed and written consent
* Patients with platelet count more than 30.000/mm3

Exclusion Criteria:

* Current alcohol consumption

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Estimated)
Dates: Start 2016-01; Primary Completion 2017-07 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
All cause mortality | one year

CONTACTS AND LOCATIONS:
Overall Officials: Murat Kantarcioglu, M.D., Study Chair — Gulhane Military Medical Academy, Department of Gastroenterology
Locations (1):
- Gulhane Military Medical Academy, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Kantarcioglu M, Demirci H, Avcu F, Karslioglu Y, Babayigit MA, Karaman B, Ozturk K, Gurel H, Akdogan Kayhan M, Kacar S, Kubar A, Oksuzoglu G, Ural AU, Bagci S. Efficacy of autologous mesenchymal stem cell transplantation in patients with liver cirrhosis. Turk J Gastroenterol. 2015 May;26(3):244-50. doi: 10.5152/tjg.2015.0074. PMID 26006200
- [Result] Kantarcioglu M, Caliskan B, Demirci H, Karacalioglu O, Kekilli M, Polat Z, Gunal A, Akinci M, Uysal C, Eksert S, Gurel H, Celebi G, Avcu F, Ural AU, Bagci S. The efficacy of mesenchymal stem cell transplantation in caustic esophagus injury: an experimental study. Stem Cells Int. 2014;2014:939674. doi: 10.1155/2014/939674. Epub 2014 May 4. PMID 24876849